CLINICAL TRIAL: NCT02056613
Title: Collection of Blood From Healthy Volunteers and Clinical Research Subjects for the Production of Clinical Grade Induced Pluripotent Stem Cell (iPSC) Products
Brief Title: Blood Collection From Healthy Volunteers and Patients for the Production of Clinical Grade Induced Pluripotent Stem Cell (iPSC) Products
Status: Withdrawn | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 140057; 14-CC-0057
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11-01

CONDITIONS: Induced Pluripotent Stem Cells
Keywords: Blood Donation; Tissue Procurement; Cellular Therapies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Pluripotent stem cells are cells that can be converted to any type of cell (muscle, nerve, liver, etc.). Researchers are collecting blood samples to develop way to make a special cell product called induced pluripotent stem cells (iPSCs). iPSCs may be used to repair or replace organs and tissues, produce blood and immune cells for transfusion, or correct inherited immune and blood diseases. iPSCs can be made from many kinds samples, such as skin, blood, or hair. This is different from embryonic stem cells, which can only be derived from embryos.

Objectives:

- To develop new methods to make iPSCs; to identify better ways to collect, produce, and grow them; and to make an iPSC bank.

Eligibility:

- Healthy adults and adults already in a treatment protocol who have a medical condition that could be treated with iPSCs.

Design:

* All participants will be screened with questionnaire, physical exam, and blood and HIV tests.
* All participants:
* Will donate 4 tablespoons of blood. It will be taken by needle from a vein in their arm.
* Participants already in another protocol:
* Will have their blood collected, separated in a lab, and iPSCs grown in large numbers. Some may have their sample given back to them as a treatment.
* Samples will be kept in the study up to 5 years or until a participant withdraws from the study or becomes ineligible to participate, or the study is closed. If participants have not withdrawn their consent, they may be contacted in the future to donate again.

DETAILED DESCRIPTION:
Induced pluripotent stem cells (iPSCs) can be produced from small quantities of blood. Clinical protocols to treat several diseases using iPSCs or cells derived from iPSCs are being developed by intramural investigators, i.e., investigators in National Institute of Allergy and Infectious Diseases (NIAID) and National Eye Institute (NEI). This clinical protocol will allow personnel in the Cell Processing Service (CPS) of the Department of Transfusion Medicine (DTM) to collect blood from healthy donors or patients with diseases targeted in IRB-approved treatment protocols to manufacture iPSCs or iPSC derived products to support these intramural investigators. CPS DTM will submit a Drug Master File (DMF) to the US Food and Drug Administration (FDA) for the manufacture and testing of these products. When iPSCs are used clinically in some cases the donors will be the recipients of the iPSCs, or the ex vivo expanded and differentiated iPSCs (autologous therapy). In other cases, healthy subjects will serve as donors of the blood used as starting material for manufacturing iPSCs (allogeneic therapy) where no matching of HLA or other antigens is required between the healthy blood donor and the iPSC recipient. While methods to produce and expand iPSCs have been described, they must be modified periodically to meet changing Good Manufacturing Practices (GMP) requirements for manufacturing clinical cell and gene therapies, therefore peripheral blood for iPSCs from normal donors is needed for research and development.

ELIGIBILITY:
* INCLUSION CRITERIA RELATED OR THIRD PARTY DONORS (ALLOGENEIC CELLS, INCLUDING RESEARCH DONORS) AND AUTOLOGOUS DONORS

Subjects who meet ALL of the following criteria will be considered for enrollment into this study:

1. Be greater than or equal to 18 years of age, as of the date of enrollment. There is no upper age limit for donor enrollment.
2. Able to provide informed consent.
3. Meets the donation requirements established by AABB and FDA for allogeneic or autologous use with the exception of hemoglobin/hematocrit.

SUBJECT EXCLUSION CRITERIA ALLOGENEIC DONORS

Subjects who meet ANY of the following criteria will be excluded from participation in this study as a third party donor or research volunteer:

1. Medical history that includes any of the following, as per AABB or FDA requirements for allogeneic use:

   * Thrombocytopenia or other blood dyscrasias
   * Bleeding diathesis
   * Antibiotic use within the prior 48 hours
   * History of cancer
   * History of exposure to transfusion transmitted diseases including HIV and hepatitis B and C as defined by the Standards for Blood Banking and Transfusion Services, AABB.
   * Travel to an area where malaria is endemic as defined by the CDC (www.cdc.gov/travel).
   * At risk for the possible transmission of Creutzfeldt-Jakob Disease (CJD) and Variant Creutzfeldt-Jakob Disease (vCJD) as described in the FDA Guidance for Industry, January 9, 2002, Revised Preventive Measures to Reduce the Possible Risk of Transfusion of Creutzfeldt-Jakob Disease (CJD) and Variant Creutzfeldt-Jakob Disease (vCJD) by Blood and Blood Products
2. Febr le (temperature >38 (Infinite)C)
3. Hemoglobin level

   * African American women <11.5 grams/dL
   * Other women <12.0 grams/dL
   * Men <12.5 grams/dL
4. HCT

   * African American women <34%
   * Other women <36%
   * Men <38%
5. Platelets <150 times 103/microL
6. Absolute neutrophil count <1.0 times 103/microL
7. Positive tests for blood borne pathogens (as required by the Standards for Blood Banks and Transfusion Services, AABB. The currently required tests include anti-HIV1/2, anti-HCV, anti-HBc, Anti-HTLV I/II, anti-T. Cruzi, HBsAg, syphilis, and molecular testing for West Nile virus, HCV, HBV, and HIV-1).

SUBJECT EXCLUSION CRITERIA AUTOLOGOUS DONORS

Subjects who meet ANY of the following criteria will be excluded from participation in this study:

1. Positive tests for anti-HIV1/2, anti-HCV, or HBsAg
2. Does not meet criteria established by the NIH IRB-approved treatment protocol for administration of iPSCs, as created by the protocol PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02-05; Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
collection of blood samples for production of iPSCs or iPSV-derived therapy products | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: David F Stroncek, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)

REFERENCES:
- [Background] Takahashi K, Yamanaka S. Induction of pluripotent stem cells from mouse embryonic and adult fibroblast cultures by defined factors. Cell. 2006 Aug 25;126(4):663-76. doi: 10.1016/j.cell.2006.07.024. Epub 2006 Aug 10. PMID 16904174
- [Background] Mostoslavsky G. Concise review: The magic act of generating induced pluripotent stem cells: many rabbits in the hat. Stem Cells. 2012 Jan;30(1):28-32. doi: 10.1002/stem.742. PMID 21948613
- [Background] Somers A, Jean JC, Sommer CA, Omari A, Ford CC, Mills JA, Ying L, Sommer AG, Jean JM, Smith BW, Lafyatis R, Demierre MF, Weiss DJ, French DL, Gadue P, Murphy GJ, Mostoslavsky G, Kotton DN. Generation of transgene-free lung disease-specific human induced pluripotent stem cells using a single excisable lentiviral stem cell cassette. Stem Cells. 2010 Oct;28(10):1728-40. doi: 10.1002/stem.495. PMID 20715179